CLINICAL TRIAL: NCT06080802
Title: The Effect of Addition of Metformin to SGLT2 In Diabetic Patients With Heart Failure With Preserved Ejection Fraction
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: October University for Modern Sciences and Arts (Other)
Collaborators: clinical research unit, El-sheikh zayed specialized hospital - Egyptian Ministry of health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C1/HEC1/2023PD
Record Dates: First submitted 2023-10-08; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Diabete Type 2
Keywords: metformin; SGLTi; HFpEF
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control(SGLT2i/ARBs/MRA/ +/- diuretics). (No Intervention): Lifestyle counseling plus standard evidence-based therapy for HFpEF (SGLT2i/ARBs/MRA/ +/- diuretics).
- intervention (Experimental): Lifestyle counseling plus standard evidence-based therapy for HFpEF (SGLT2i/ARBs/MRA/ +/- diuretics)+ metformin
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — The intervention will consist in giving metformin starting with 500 mg once daily 1 gm daily (at breakfast) during the first week; if well tolerated, the dose was progressively increased to 500 mg twice daily (at breakfast and dinner) during week 2, to 1000 mg at breakfast and 500 mg at dinner during week 3, in order to reach the target dose of 1000 mg twice daily (at breakfast and dinner) during the rest of the follow-up. Patients will be followed up by telephone call 2 weeks intervals during the study period 5 SGL-2 will be prescribed to group 1 after diagnosis with HFpEF while group 2 will have SGL-2 and Metformin
  Arms: intervention

SUMMARY:
a prospective open-label, randomized controlled study to evaluate the efficacy of the addition of metformin to SGLT2 in diabetic patient with preserved ejection fraction

DETAILED DESCRIPTION:
Regardless of the benefits noted with SGLT2is, metformin is recommended as first-line therapy for glycemic control in individuals with T2DM and HF, including HFpEF, with estimated glomerular filtration rates (eGFRs) ≥30 mL/min/1.73 m2. This is based on the demonstrated experience with long-term use; its safety, low cost, and low side effect profile; as well as observational (not clinical trial) data suggesting a 20% relative risk reduction in mortality in individuals with HF, including HFpEF.

Nevertheless, it is worth mentioning that Metformin is a common anti-diabetic drug with both systemic and cardioprotective benefits in addition to its hypoglycaemic effect. At the cellular level metformin activates adenosine monophosphate-activated protein kinase (AMPK) an important regulator of several metabolic pathways resulting in enhanced glucose utilisation, reduction of protein synthesis and improvement of mitochondrial function. Furthermore, metformin has been shown to reduce collagen accumulation and potentially reduce LV hypertrophy and improve diastolic function in the diabetic myocardium. The cardio protection afforded by metformin treatment seems to result from interference with TGF-beta signaling pathway and activation of the AMP-kinase signaling cascade. A recent systematic review and meta regression analysis have shown that metformin treatment was associated with a reduction in mortality in patients with HFpEF. In addition, treatment with metformin of non-diabetic metabolic syndrome patients with diastolic dysfunction, on top of lifestyle counseling, was associated with improved diastolic function.

Nevertheless, a recent met analysis showed that initial SGLT2 inhibitor/metformin combination therapy has glycaemic and weight benefits compared with either agent alone and appears relatively safe. High dose SGLT2 inhibitor/metformin combination therapy appears to have modest weight, but no glycaemic benefits compared with the low dose combination therapy.

based on that we our aim is to evaluate the efficacy of the addition of metformin to SGLT2 in diabetic patient with preserved ejection fraction

ELIGIBILITY:
Inclusion Criteria:

Age of 40 years to 74 years. HFpEF (≥ 50%) Written informed consent of the subject to participate in the study. New York Heart Association functional class I-IV. Diabetic patients SGL-2 naive. Newly diagnosed heart failure of preserved ejection fraction

Exclusion Criteria:

Patients with heart failure with reduced ejection fraction (< 40%) Age less than 40 and more than 74 GFR < 30 mL/min A1c > 9 Known allergy to metformin End- stage liver disease Cancer Pregnancy or lactation

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Hospitalization rate | baseline, 3 and 6 months
  Hospitalization rate
HRQOL using Minnesota Living with Heart Failure Questionnaire for quality-of-life evaluation (MLFHQ) | baseline, 3 and 6 months
  HRQOL using Minnesota Living with Heart Failure Questionnaire for quality-of-life evaluation (MLFHQ)

SECONDARY OUTCOMES:
The change in the mean early diastolic mitral annular velocity (mean e'), at 3 and 6 months | baseline, 3 and 6 months
  The change in the mean early diastolic mitral annular velocity (mean e'), at 3 and 6 months
adverse drug effects | baseline, 3 and 6 months
  adverse drugs effects
Change in N-terminal pro-BNP (NT-proBNP) | baseline, 3 and 6 months
  Change in N-terminal pro-BNP (NT-proBNP)
Neutrophil/lymphocyte ratio -AMPK pathway | baseline, 3 and 6 months
  Neutrophil/lymphocyte ratio
  -AMPK pathway
Inflammatory and oxidative stress | baseline, 3 and 6 months
  Inflammatory and oxidative stress
Change in body weight | baseline, 3 , 6 months
  Change in body weight

CONTACTS AND LOCATIONS:
Overall Officials: sara M eladawy, Study Director — MSA university; Mai abdelhafez, PhD, Study Chair — MSA university
Locations (1):
- clinical research uint- El-sheikh zayed specialized hospital SMC- Egyptian Ministry of health, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ElSayed NA, Aleppo G, Aroda VR, Bannuru RR, Brown FM, Bruemmer D, Collins BS, Hilliard ME, Isaacs D, Johnson EL, Kahan S, Khunti K, Leon J, Lyons SK, Perry ML, Prahalad P, Pratley RE, Seley JJ, Stanton RC, Gabbay RA, on behalf of the American Diabetes Association. 9. Pharmacologic Approaches to Glycemic Treatment: Standards of Care in Diabetes-2023. Diabetes Care. 2023 Jan 1;46(Suppl 1):S140-S157. doi: 10.2337/dc23-S009. PMID 36507650
- [Background] Kittleson MM, Panjrath GS, Amancherla K, Davis LL, Deswal A, Dixon DL, Januzzi JL Jr, Yancy CW. 2023 ACC Expert Consensus Decision Pathway on Management of Heart Failure With Preserved Ejection Fraction: A Report of the American College of Cardiology Solution Set Oversight Committee. J Am Coll Cardiol. 2023 May 9;81(18):1835-1878. doi: 10.1016/j.jacc.2023.03.393. Epub 2023 Apr 19. No abstract available. PMID 37137593